CLINICAL TRIAL: NCT01396135
Title: A Phase 1, Randomized, Subject- And Investigator-blind, Sponsor-open, Placebo-controlled, Single- And Multiple-dose Study To Investigate The Pharmacokinetics, Safety And Tolerability Of Cp-601,927 In Healthy Japanese Subjects
Brief Title: A Phase 1 Study To Investigate The Pharmacokinetics, Safety And Tolerability Of CP-601,927 In Healthy Japanese Subjects
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: A3331019
Record Dates: First submitted 2011-07-14; First posted 2011-07-18 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Healthy
Keywords: Phase 1; Pharmacokinetics; Healthy; Japanese; Non-smokers; Major Depressive Disorder; CP-601; 927
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single dosing (Experimental): Single doses of CP-601,927 (1, 2 or 3 mg) or placebo
  Interventions: Drug: CP-601,927; Drug: Placebo
- Multiple dosing (Experimental): Multiple doses of CP-601,927 (2 mg BID, 4mg/day) or placebo
  Interventions: Drug: CP-601,927; Drug: Placebo

INTERVENTIONS:
Drug: CP-601,927 — Single dose of 1 mg CP-601,927 given as oral 1 mg tablets
  Arms: Single dosing
Drug: CP-601,927 — Single dose of 2 mg CP-601,927 given as oral 1 mg tablets
  Arms: Single dosing
Drug: CP-601,927 — Single dose of 3 mg CP-601,927 given as oral 1 mg tablets
  Arms: Single dosing
Drug: Placebo — Single dose of placebo given as a matching number of oral tablets
  Arms: Single dosing
Drug: CP-601,927 — Multiple doses of CP-601,927 given as 2 mg BID (4 mg/day) as oral 1 mg tablets for 7 days
  Arms: Multiple dosing
Drug: Placebo — Multiple doses of placebo given as a matching number of oral tablets
  Arms: Multiple dosing

SUMMARY:
This Phase 1 study is the first clinical trial to be conducted in Japanese subjects. The pharmacokinetics, safety and tolerability of single and multiple doses of CP-601,927 will be evaluated in Japanese, healthy, non-smoking subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female Japanese subjects between the ages of 18 and 55 years, inclusive.
* Japanese defined as being able to document that all 4 grandparents were Japanese and were born in Japan.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Females of childbearing potential.
* Subjects with regular (daily or weekly) use of tobacco products or nicotine currently or within the past 6 months. Subjects with urine cotinine concentrations >100 ng/mL at any time during the study will be excluded.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-08-26 (Actual); Primary Completion 2011-10-29 (Estimated); Study Completion 2011-10-29 (Estimated)

PRIMARY OUTCOMES:
Cmax, AUClast, AUC0-12, Tmax and as data permit AUCinf, t1/2, CL/F, Vd/F after single dose of 1 mg CP-601,927 | 0,0.5,1,2,4,6,8,12,14,16,24,36,48 hours post-dose
Cmax, AUClast, AUC0-12, Tmax and as data permit AUCinf, t1/2, CL/F, Vd/F after single dose of 2 mg CP-601,927 | 0,0.5,1,2,4,6,8,12,14,16,24,36,48 hours post-dose
Cmax, AUClast, AUC0-12, Tmax and as data permit AUCinf, t1/2, CL/F, Vd/F after single dose of 3 mg CP-601,927 | 0,0.5,1,2,4,6,8,12,14,16,24,36,48 hours post-dose
Ctrough, Cmax, AUC0-12, Tmax and as data permit t1/2, CL/F and Rac (accumulation ratio) based on Cmax and AUC0-12 after multiple doses of CP-601,927 given as 2 mg BID (4mg/day) for 7 days | Day1-7
Suicidality assessment after single dose of 1 mg CP-601,927 | Day 0, 0 and 2 hours post-dose
Suicidality assessment after single dose of 2 mg CP-601,927 | Day 0, 0 and 2 hours post-dose
Suicidality assessment after single dose of 3 mg CP-601,927 | Day 0, 0 and 2 hours post-dose
Suicidality assessment after multiple doses of CP-601,927 given as 2 mg BID (4mg/day) for 7 days | Day1-7

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3331019&StudyName=A%20Phase%201%20Study%20To%20Investigate%20The%20Pharmacokinetics%2C%20Safety%20And%20Tolerability%20Of%20CP-601%2C927%20In%20Healthy%20Japanese%20Subjects